CLINICAL TRIAL: NCT02013063
Title: Accuracy and Cost-Effectiveness of Dynamic Contrast Enhanced Computed Tomography in the Characterisation of Solitary Pulmonary Nodules
Brief Title: Single Pulmonary Nodule Investigation
Acronym: SPUtNIk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other); Brighton and Sussex University Hospitals NHS Trust (Other); University College London Hospitals (Other); Oxford University Hospitals NHS Trust (Other); Papworth Hospital NHS Foundation Trust (Other Government); The Leeds Teaching Hospitals NHS Trust (Other); Manchester University NHS Foundation Trust (Other Government); East and North Hertfordshire NHS Trust (Other Government); NHS Grampian (Other Government); NHS Greater Glasgow and Clyde (Other); Western Sussex Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHM RAD0030; ISRCTN30784948 (Other: ISRCTN); project number 09/22/117 (Other Grant/Funding Number: NIHR-HTA)
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Malignant Neoplasm of Lung
Keywords: Single Pulmonary Nodule; SPN; Lung cancer; Diagnostic; Computed Tomography; CT scan; FDG-PET scan; Dynamic CT scan; DCE-CT scan; Dynamic contrast enhanced CT scan; soft tissue solitary dominant; ≥ 8mm and ≤30mm
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A small proportion of patients with lung cancer present with a solitary pulmonary nodule (SPN). This is an important group of patients because if it is lung cancer, presentation as a SPN represents early disease, which following surgery has a high 5 year survival rate. However as not all SPNs are lung cancer it would be unethical to biopsy every case. Clinical guidelines recommend that SPNs should undergo an initial (FDG)-PET/CT scan, which may give more information about the SPN and may indicate if it is likely to be lung cancer. However in many cases it does not and current practice is to monitor the SPN with a series of CT scans over 2 years to look for changes or growth which may/ but not always indicate lung cancer. If no changes are observed over 2 years the SPN is considered not lung cancer. This is both expensive for the National Health Service (NHS) and worrying for the patient in terms of monitoring CT costs and delayed treatment due to length of time to diagnosis.

This study examines the diagnostic capacity of using a different CT scan. Dynamic Contrast Enhanced -CT(DCE-CT). DCE-CT and FDG-PET/CT scans give different information about the SPN and the investigators will look to see if information from either scan or combined information from both scans may be better in the diagnosis of early stage lung cancer. The investigators will also undertake a review of previous studies that have used these scans and use data from both the review and the trial to look at the cost effectiveness of using DCE-CT in the diagnosis of SPN.

The trial will recruit 375 people who have a SPN detected by a normal CT scan which requires a FDG-PET/CT scan. In addition they will receive a DCE-CT scan either on the same day or within three weeks of the FDG-PET/CT scan. This is the only extra procedure that will take place to normal NHS care, however we will collect clinical and outcome data over the next two years.

The study is coordinated by Southampton University clinical trials unit. Recruitment between January 2013 - April 2016, from up to 14 UK sites. Data analysis and conclusions are expected by the end of 2018.

The study is funded by the NIHR-HTA

DETAILED DESCRIPTION:
Indication: Lung Cancer

Primary Objectives:

* To determine with high precision, the diagnostic performances of DCE-CT and 18FDG-PET/CT in the NHS for the characterisation of solitary pulmonary nodules (SPNs).
* To use decision analytic modelling to assess the likely costs and health outcomes resulting from incorporation of DCE-CT into management strategies for patients with SPNs.

Secondary Objectives:

* To assess, within an NHS setting, the incremental value of incorporating the CT appearances of a SPN into the interpretation of integrated PET/CT examinations.
* To assess whether combining DCE-CT with 18FDG-PET/CT is more accurate and/or cost-effective, in the characterisation of SPNs, than either test used alone or in series.
* To document the nature and incidence of incidental extra-thoracic findings on 18FDG-PET/CT undertaken for the characterisation of SPNs and model their impact on cost-effectiveness.

Rationale:

A small proportion of patients with lung cancer present with a solitary pulmonary nodule (SPN) on diagnostic imaging tests. This is an important group of patients because presentation as a SPN represents early disease with high 5 year survival rates following surgical resection. However, not all SPNs are due to lung cancer and the accurate characterisation of SPNs for diagnosis of early stage lung cancer is a diagnostic challenge with significant associated health costs.

Widely adopted clinical guidelines for the subsequent investigation of SPNs recommend serial CT scans to look for subsequent growth with biopsy to confirm diagnosis. UK, National Institute for Health and Clinical Excellence (NICE) guidelines recommend 18FDG-PET for the assessment of SPN in cases where a biopsy is not possible or has failed.

DCE-CT and 18FDG-PET scans give different information about the SPN. Information from either scan or combined information from both scans may be better in the diagnosis of early stage lung cancer.

Trial Design: Prospective Observational

Sample size: 375

Non-CTIMP:Non interventional trial

Concomitant Therapy: As per local practice

Primary Trial Endpoints:

Primary outcome measures will include diagnostic test characteristics (sensitivity, specificity, accuracy) for 18FDG-PET/CT and DCE-CT in relation to a subsequent clinical diagnosis of lung cancer. The outcome measures used in the economic model will include accuracy, estimated life expectancy, and quality adjusted life years (QALYs). Costs will be estimated from an NHS perspective. Incremental cost-effectiveness ratios will compare management strategies with DCE-CT to strategies without DCE-CT.

Secondary Trial Endpoints:

Secondary outcome measures will include diagnostic test characteristics for 18FDG-PET/CT with incorporation of CT appearances and combined DCE-CT/18FDG-PET. The incidence of incidental extra-thoracic findings on 18FDG-PET/CT, subsequent investigations and costs will also be determined.

Total Number of Sites: up to 14

ELIGIBILITY:
Inclusion Criteria:

* A soft tissue solitary dominant pulmonary nodule of ≥ 8mm and ≤30mm on axial plane

  * Measured on lung window using conventional CT scan
  * No other ancillary evidence strongly indicative of malignancy (e.g. distant metastases or unequivocal local invasion).
* If clinicians and reporting radiologists believe the patient is being treated as having a single pulmonary nodule and there are other small lesions <4mm that would normally be disregarded, the patient should be included in the trial.
* Nodules already under surveillance can be included provided they have a recent or scheduled FDG-PET/CT18 years of age or over at time of providing consent
* Able and willing to consent to study

Exclusion Criteria:

* Pregnancy
* History of malignancy within the past 2 years
* Confirmed aetiology of the nodule at the time of qualifying CT scan - As this is a diagnostic study, should the aetiology of the nodule be confirmed by investigation such as FDG-PET/CT or bronchoscopy prior to consent the patient remains eligible as the intention to include is made on the analysis of the qualifying CT scan.
* Biopsy of nodule prior to DCE-CT scan
* Contra-indication to potential radiotherapy or surgery
* Contra indication to scans (assessed by local procedures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital Chest Clinics PET referal centres
Sampling Method: Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2012-08; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of DCE-CT scans and FDG-PET scans to diagnose early lung cancer in SPN | 2 years
  Primary outcome measures will include diagnostic test characteristics (sensitivity, specificity, accuracy) for 18FDG-PET/CT and DCE-CT in relation to a subsequent clinical diagnosis of lung cancer.
cost effectiveness of using DCE-CT scans in the diagnosis of early lung cancer in SPN | 2 years
  The outcome measures used in the economic model will include accuracy, estimated life expectancy, and quality adjusted life years (QALYs). Costs will be estimated from an NHS perspective. Incremental cost-effectiveness ratios will compare management strategies with DCE-CT to strategies without DCE-CT.

SECONDARY OUTCOMES:
Effectiveness of DCE-CT scans combined with FDG-PET scans to diagnose early lung cancer in SPN | 2 years
  Diagnostic test characteristics combined DCE-CT/18FDG-PET in relation to a subsequent clinical diagnosis of lung cancer.
Effectiveness of using analysis of the CT image from the FDG-PET/CT in conjunction with data from the FDG incorporation to diagnose early lung cancer in SPN | 2 years
  Diagnostic test characteristics for 18FDG-PET/CT with incorporation of CT appearances in relation to a subsequent clinical diagnosis of lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Steve George, MD,FRCP, Principal Investigator — University of Southampton
Locations (9):
- United Kingdom (9):
  - Southampton University Hospitals Nhs Trust, Southampton, Hampshire
  - Western Sussex Hospitals NHS Foundation Trust, Worthing, Sussex
  - NHS Grampian, Aberdeen
  - Brighton and Sussex University Hospitals Nhs Trust, Brighton
  - Papworth Hospital Nhs Foundation Trust, Cambridge
  - NHS Greater Glasgow and Clyde, Glasgow
  - Leeds Teaching Hospitals Nhs Trust, Leeds
  - University College London Hospitals Nhs Foundation Trust, London
  - University Hospital of South Manchester Nhs Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No
there is no plan to share individual patient data

REFERENCES:
- [Derived] Weir-McCall JR, Debruyn E, Harris S, Qureshi NR, Rintoul RC, Gleeson FV, Gilbert FJ; SPUtNIk Investigators. Diagnostic Accuracy of a Convolutional Neural Network Assessment of Solitary Pulmonary Nodules Compared With PET With CT Imaging and Dynamic Contrast-Enhanced CT Imaging Using Unenhanced and Contrast-Enhanced CT Imaging. Chest. 2023 Feb;163(2):444-454. doi: 10.1016/j.chest.2022.08.2227. Epub 2022 Sep 8. PMID 36087795
- [Derived] Gilbert FJ, Harris S, Miles KA, Weir-McCall JR, Qureshi NR, Rintoul RC, Dizdarevic S, Pike L, Sinclair D, Shah A, Eaton R, Clegg A, Benedetto V, Hill JE, Cook A, Tzelis D, Vale L, Brindle L, Madden J, Cozens K, Little LA, Eichhorst K, Moate P, McClement C, Peebles C, Banerjee A, Han S, Poon FW, Groves AM, Kurban L, Frew AJ, Callister ME, Crosbie P, Gleeson FV, Karunasaagarar K, Kankam O, George S. Dynamic contrast-enhanced CT compared with positron emission tomography CT to characterise solitary pulmonary nodules: the SPUtNIk diagnostic accuracy study and economic modelling. Health Technol Assess. 2022 Mar;26(17):1-180. doi: 10.3310/WCEI8321. PMID 35289267
- [Derived] Gilbert FJ, Harris S, Miles KA, Weir-McCall JR, Qureshi NR, Rintoul RC, Dizdarevic S, Pike L, Sinclair D, Shah A, Eaton R, Jones J, Clegg A, Benedetto V, Hill J, Cook A, Tzelis D, Vale L, Brindle L, Madden J, Cozens K, Little L, Eichhorst K, Moate P, McClement C, Peebles C, Banerjee A, Han S, Poon FW, Groves AM, Kurban L, Frew A, Callister MEJ, Crosbie PA, Gleeson FV, Karunasaagarar K, Kankam O, George S. Comparative accuracy and cost-effectiveness of dynamic contrast-enhanced CT and positron emission tomography in the characterisation of solitary pulmonary nodules. Thorax. 2022 Oct;77(10):988-996. doi: 10.1136/thoraxjnl-2021-216948. Epub 2021 Dec 9. PMID 34887348
- [Derived] Weir-McCall JR, Harris S, Miles KA, Qureshi NR, Rintoul RC, Dizdarevic S, Pike L, Cheow HK, Gilbert FJ; SPUtNIk investigators. Impact of solitary pulmonary nodule size on qualitative and quantitative assessment using 18F-fluorodeoxyglucose PET/CT: the SPUTNIK trial. Eur J Nucl Med Mol Imaging. 2021 May;48(5):1560-1569. doi: 10.1007/s00259-020-05089-y. Epub 2020 Nov 1. PMID 33130961